CLINICAL TRIAL: NCT05454631
Title: Satisfaction Survey on the Tolerability of Surgical Masks for Protection Against the Spread of SARS-CoV2 in Patients With Chronic Respiratory Diseases
Brief Title: Tolerance of Surgical Masks in Chronic Respiratory Diseases
Acronym: TOLMASK
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APHP220201
Record Dates: First submitted 2022-07-07; First posted 2022-07-12 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: breathlessness; face masks; COVID-19; COPD; pulmonary rehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea; COVID-19

STUDY DESIGN:
Masking Description: not everyone involved in the research (patients, investigators, caregivers, and statistical analysis stakeholders) will know which mask the patient is using at which time.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patient present at the respiratory SSR department of the Pitié-Salpêtrière hospital (Experimental): All the participants will evaluate 5 different types of surgical mask, in random order.
  Interventions: Device: surgical mask (5 different types)

INTERVENTIONS:
Device: surgical mask (5 different types) — All the participants will wear 5 different types of surgical mask, in random order.

SUMMARY:
The study is conducted in the context of the COVID-19 pandemic in general, and more specifically in the context of the evaluation of the use of protective masks as a barrier to the spread of the virus. The wearing of masks is one of the recommended barrier measures to limit the spread of the SARS-CoV-2 virus responsible for COVID-19. It is recommended in all circumstances, and mandatory in some. Regardless of the type of mask used (noting that the so-called "surgical" masks are by far the most common), there are various disadvantages associated with wearing them. Dyspnoea (unpleasant or upsetting perception of respiratory activity) is one of these disadvantages. It can lead to reluctance to wear the mask, or to the adoption of inappropriate practices that reduce its effectiveness. This "side effect" of the mask is more pronounced in patients with underlying respiratory diseases. However, not all mask designs are equivalent in terms of their physical properties, which can theoretically generate varying levels of dyspnoea. It is therefore important to determine which mask designs are more or less dyspnogenic, in order to guide the preferential use of certain designs in certain patient categories. The TOLMASK study (Tolerance of SARS-CoV2 Surgical Masks in Patients with Chronic Respiratory Diseases) is a prospective, randomised, triple-blind, single-centre study comparing several surgical masks in a crossover design. The primary objective of the study is to evaluate the respiratory tolerance of different surgical masks and the secondary objective is to evaluate their general tolerance.

DETAILED DESCRIPTION:
The study was conducted in the context of the COVID-19 pandemic in general, and more specifically in the context of the evaluation of the use of protective masks as a barrier to the spread of the virus. The wearing of masks is one of the recommended barrier measures to limit the spread of the SARS-CoV-2 virus responsible for COVID-19. It is recommended in all circumstances, and mandatory in some. Regardless of the type of mask used (noting that the so-called "surgical" masks are by far the most common), there are various disadvantages associated with wearing them. Dyspnoea (unpleasant or worrying perception of respiratory activity) is one of these disadvantages. It can lead to reluctance to wear the mask, or to the adoption of inappropriate practices that reduce its effectiveness. This "side effect" of the mask is more pronounced in patients with underlying respiratory diseases. However, not all mask designs are equivalent in terms of their physical properties, which can theoretically generate varying levels of dyspnoea. It is therefore important to determine which mask designs are more or less dyspnogenic, in order to guide the preferential use of certain designs in certain patient categories. The TOLMASK study (Tolerance of SARS-CoV2 Surgical Masks in Patients with Chronic Respiratory Diseases) is a prospective, randomised, triple-blind, single-centre study comparing several surgical masks in a crossover design. The primary objective of the study is to evaluate the respiratory tolerance of different surgical masks and the secondary objective is to evaluate their general tolerance.

The inclusion criteria are : 1) patient hospitalised in the respiratory and neuro-respiratory rehabilitation department of the R3S department at the Pitié-Salpêtrière Hospital (Pr Gonzalez-Bermejo); 2) patient enrolled in a respiratory rehabilitation process including exercise training on a cyclo-ergometer or treadmill; 3) hospitalisation in the respiratory rehabilitation department either post-exacerbation of COPD (usual recruitment of the department) or post-COVID (depending on the epidemic situation at the time of the study); 4) patient of age.

The criteria for non-inclusion are 1) Exercise re-training under mask ventilatory assistance; 2) Presence of a tracheotomy; 3) Psychiatric disorders (at the discretion of the referring physician); 4) Insufficient command of the French language; 5) Refusal to participate in the study.

50 patients will be included, over a period of 4 months. The duration of participation is 5 days.

ELIGIBILITY:
Inclusion Criteria:

* Patient hospitalised in the respiratory and neuro-respiratory SSR service of the R3S department at the Pitié-Salpêtrière Hospital (Pr Gonzalez-Bermejo)
* Patient enrolled in a respiratory rehabilitation process including exercise training on a cyclo-ergometer or treadmill
* Hospitalization in respiratory rehabilitation unit either in post-exacerbation of COPD
* age over 18

Exclusion Criteria:

* Exercise training under mask ventilation support
* Presence of a tracheostomy
* Psychiatric disorders (at the discretion of the referring physician)
* Insufficient command of the French language
* Refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-02-06 (Actual); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
affective dimension of dyspnea | immediately after a rehabilitation session
  Intensity of the sensory dimension of respiratory discomfort attributed to wearing the mask during exercise training, assessed on an 11-point ordinal scale (from "0, the mask caused no particular respiratory sensation" to "10, the mask caused a respiratory sensation as intense as I can imagine")

SECONDARY OUTCOMES:
sensory dimension of dyspnea | immediately after a rehabilitation session
  Intensity of the sensory dimension of respiratory discomfort attributed to wearing the mask during exercise training, assessed on an 11-point ordinal scale (from "0, the mask caused no particular respiratory sensation" to "10, the mask caused a respiratory sensation as intense as I can imagine")
relief | immediately after a rehabilitation session
  Intensity of relief on mask removal, rated on an 11-point ordinal scale (from "0, mask removal caused no relief" to "10, mask removal caused absolute relief")
MDP (Multidimensional Dyspnea Profile) | immediately after a rehabilitation session
  Response to the Multidimensional Dyspnea Profile questionnaire (French version) The Multidimensional Dyspnoea Profile (MDP) consists of eleven 0-10 numerical rating scales describing the unpleasantness of dyspnea (A1, maximum score of 10), its sensory qualities (5 items [SQ], maximum 50), and its emotional qualities (5 items [A2], maximum 50).
general comfort | immediately after a rehabilitation session
  Overall comfort of the mask tested, rated on an 11-point ordinal scale (from "0, this mask is horribly uncomfortable", to "10, this mask is perfectly comfortable").
choice | immediately after a rehabilitation session
  Overall comfort of the mask tested, rated on Choice and ranking of 5 mask disadvantages from a list of 15 In addition, at the end of the study, patients will be asked to indicate which of the masks tested they preferred.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas SIMILOWSKI, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Département R3S, Hôpital Pitié-Salpêtrière, Paris, France

REFERENCES:
- [Background] Serresse L, Simon-Tillaux N, Decavele M, Gay F, Nion N, Lavault S, Guerder A, Chatelet A, Dabi F, Demoule A, Morelot-Panzini C, Moricot C, Similowski T. Lifting dyspnoea invisibility: COVID-19 face masks, the experience of breathing discomfort, and improved lung health perception - a French nationwide survey. Eur Respir J. 2022 Mar 31;59(3):2101459. doi: 10.1183/13993003.01459-2021. Print 2022 Mar. PMID 34475232